CLINICAL TRIAL: NCT00063453
Title: The Respiratory Ancillary Study (RAS) to SELECT
Brief Title: Supplemental Selenium and Vitamin E and Pulmonary Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 151; R01HL071022 (NIH); NCT00241865 (obsolete NCT alias); NCT00782678 (obsolete NCT alias)
Record Dates: First submitted 2003-06-26; First posted 2003-06-30 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Diseases; Lung Diseases, Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive | interventions — Vitamin E; Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin E and selenium placebo (Experimental): Vitamin E alone
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Selenium placebo
- Selenium and vitamin E placebo (Experimental): Selenium alone
  Interventions: Dietary Supplement: Selenium; Dietary Supplement: Vitamin E placebo
- Vitamin E and selenium (Experimental): Vitamin E and selenium combined
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Selenium
- vitamin E Placebo and Selenium placebo (Placebo Comparator): Double placebo
  Interventions: Dietary Supplement: Vitamin E placebo; Dietary Supplement: Selenium placebo

INTERVENTIONS:
Dietary Supplement: Vitamin E — vitamin E (400 IU/day all rac-α-tocopheryl acetate)
  Other Names: all rac-α-tocopheryl acetate
  Arms: Vitamin E and selenium; Vitamin E and selenium placebo
Dietary Supplement: Selenium — selenium (200 μg/d L-selenomethionine)
  Other Names: L-selenomethionine
  Arms: Selenium and vitamin E placebo; Vitamin E and selenium
Dietary Supplement: Vitamin E placebo — placebo
  Other Names: Placebo
  Arms: Selenium and vitamin E placebo; vitamin E Placebo and Selenium placebo
Dietary Supplement: Selenium placebo — placebo
  Other Names: placebo
  Arms: Vitamin E and selenium placebo; vitamin E Placebo and Selenium placebo

SUMMARY:
To test whether supplementation with selenium and/or vitamin E affects pulmonary function.

DETAILED DESCRIPTION:
BACKGROUND:

There is compelling evidence from observational epidemiologic studies that intakes of nutrients with antioxidant properties are associated with reduced risks of chronic obstructive disease (COPD) and increased lung function. This study is ancillary to the multisite Selenium and Vitamin E Cancer Prevention Trial (SELECT), a 4-arm placebo-controlled, double-blinded randomized trial in 35,000 men testing whether daily supplementation with vitamin E (400mg alpha-tocopherol), selenium (200 micrograms selenomethionine) or both vitamin E and selenium can prevent prostate cancer.

DESIGN NARRATIVE:

This study is ancillary to the multisite Selenium and Vitamin E Cancer Prevention Trial (SELECT), a 4-arm placebo-controlled, double-blinded randomized trial in 35,000 men testing whether daily supplementation with vitamin E (400mg alpha-tocopherol), selenium (200 micrograms selenomethionine) or both vitamin E and selenium can prevent prostate cancer. A total of 3,000 SELECT participants will be enrolled for this respiratory ancillary study, and data collection will be extended to include pulmonary function, respiratory disease, and respiratory symptoms. Biological measures of nutrient exposure (serum vitamin E and selenium) and plasma lipids (total and high-density lipoprotein cholesterol) will be collected on all participants and oxidant burden (urinary F2-isoprostane) on a sub sample of heavy smokers and men with COPD. The primary outcome will be change over about 36 months in forced expiratory volume in the first second (FEV1). FEV1 is a valid and reliable measure of respiratory function that strongly predicts COPD and mortality. Extensive data on diet and dietary supplement use are being collected by the SELECT parent study. All specific aims examine pre-specified contrasts between the 4 arms of the SELECT randomized trial. The underlying hypothesis is that supplements will reduce the age related decline in FEV1 and thus at the 3-year follow-up FEV1, which will be tested in longitudinal and cross-sectional models. A secondary aim considers whether the effect of supplementation is greater among smokers (high burden of exogenous oxidants) who, by purposive selection of the study sites, will comprise about 25% of the sample.

ELIGIBILITY:
Eligibility criteria:

* age ≥ 55 y (≥ 50 y in African-Americans)
* serum prostate-specific antigen ≤ 4ng/mL
* no clinical evidence of prostate cancer

Exclusion criteria:

* Off both SELECT supplements

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2920 (Actual)
Dates: Start 2003-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary function over time by arm of study | Outcome is assessed at annual and bi-annual study visits, during in-person visit of participant to the study site. Over a period of about 36 to 48 months, participants are assessed between 3 and 4 times

OTHER OUTCOMES:
Effect of selenium and vitamin E supplementation on incidence of COPD | Questionnaire data on incident lung disease is assessed at annual and biannual study visits, in all SELECT participants. These questionnaire data were collected through the end of SELECT active follow-up, which was December 2010
  The incidence of COPD will be assessed in the full SELECT trial, given this ancillary study added questionnaire data to assess self-reported incidence of lung disease in the full 35,000 participants

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Cassano, PhD, Principal Investigator — Cornell University

REFERENCES:
- [Derived] Goodman PJ, Tangen CM, Darke AK, Arnold KB, Hartline J, Yee M, Anderson K, Caban-Holt A, Christen WG, Cassano PA, Lance P, Klein EA, Crowley JJ, Minasian LM, Meyskens FL. Opportunities and challenges in incorporating ancillary studies into a cancer prevention randomized clinical trial. Trials. 2016 Aug 12;17:400. doi: 10.1186/s13063-016-1524-9. PMID 27519183
- [Derived] Guertin KA, Grant RK, Arnold KB, Burwell L, Hartline J, Goodman PJ, Minasian LM, Lippman SM, Klein E, Cassano PA. Effect of long-term vitamin E and selenium supplementation on urine F2-isoprostanes, a biomarker of oxidative stress. Free Radic Biol Med. 2016 Jun;95:349-56. doi: 10.1016/j.freeradbiomed.2016.03.010. Epub 2016 Mar 22. PMID 27012420
- [Derived] Cassano PA, Guertin KA, Kristal AR, Ritchie KE, Bertoia ML, Arnold KB, Crowley JJ, Hartline J, Goodman PJ, Tangen CM, Minasian LM, Lippman SM, Klein E. A randomized controlled trial of vitamin E and selenium on rate of decline in lung function. Respir Res. 2015 Mar 11;16(1):35. doi: 10.1186/s12931-015-0195-5. PMID 25889509